CLINICAL TRIAL: NCT04198324
Title: Isthmocele After Endometrial and Non-endometrial Suturing in Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Şener Gezer, Principal Investigator, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KIA 2019/94
Record Dates: First submitted 2019-12-12; First posted 2019-12-13 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Cesarean Section; Dehiscence; Cesarean Wound; Dehiscence

STUDY DESIGN:
Intervention Model Description: Closure of the hysterotomy at the time of primary cesarean section
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Entire fold uterine closure (Active Comparator): The uterus will be sewn with full fold locked sutures that pass through myometrium and endometrium.
  Interventions: Procedure: Closure of the uterus with endometrium at the time of cesarean
- Non-endometrial uterine closure (Experimental): The uterus will be sewn with locked sutures that pass through myometrium without endometrium.
  Interventions: Procedure: Closure of the uterus without endometrium at the time of cesarean

INTERVENTIONS:
Procedure: Closure of the uterus with endometrium at the time of cesarean — Closure of the uterus at the time of primary cesarean will be performed with suturing the endometrium.
  Arms: Entire fold uterine closure
Procedure: Closure of the uterus without endometrium at the time of cesarean — Closure of the uterus at the time of primary cesarean will be performed without suturing the endometrium.
  Arms: Non-endometrial uterine closure

SUMMARY:
This study compares the effect of two techniques of uterine closure, with or without endometrial suturing on isthmocele development after cesarean section.

DETAILED DESCRIPTION:
Cesarean section is the most common surgery performed on pregnant women. Poor healing of the incision of the uterus leads to isthmocele development. Long-term morbidities associated with isthmocele are uterine scar pregnancy, uterine perforation, pelvic pain, and spotting-style bleeding after menstruation. Many factors that may affect the healing of uterine scar have been studied in the literature (i.e. Double or single-layer closure, locked or unlocked closure, uterine retroflection). Suturing complete fold of the wound lips during the closure of the uterus may cause the endometrial layer to be embedded in the myometrium and to form niche tissue. The study hypothesized that isthmocele development can be reduced by suturing without enclosing the endometrium during uterine closure.

ELIGIBILITY:
Inclusion Criteria:

* Term pregnancy (≥37 weeks of gestation)
* Singleton pregnancy
* Primary cesarean

Exclusion Criteria:

* Previous cesarean section
* Previous uterine surgery
* Multiple gestations
* Mullerian anomalies
* Active labor
* Placenta previa/accreta

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women
Enrollment: 170 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
Number of patients with isthmocele six month after cesarean section | 6 months after intervention
  Residual myometrium thickness of less then 2.5 mm with transvaginal ultrasonography
Mean myometrium thickness | 6 months after intervention
  Myometrial thickness measured at incision site with transvaginal ultrasonography

SECONDARY OUTCOMES:
Spotting | 6 months after intervention
  The rate of spotting complains of patients

CONTACTS AND LOCATIONS:
Overall Officials: Şener Gezer, M.D, Principal Investigator — Kocaeli University
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bij de Vaate AJ, van der Voet LF, Naji O, Witmer M, Veersema S, Brolmann HA, Bourne T, Huirne JA. Prevalence, potential risk factors for development and symptoms related to the presence of uterine niches following Cesarean section: systematic review. Ultrasound Obstet Gynecol. 2014 Apr;43(4):372-82. doi: 10.1002/uog.13199. PMID 23996650